CLINICAL TRIAL: NCT04722393
Title: Outcomes of Pulmonary Rehabilitation After Lung Resection in Patients With Non-Small Cell Lung Cancer
Brief Title: Lung Resection and Pulmonary Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Ilknur Naz, Assoc. Prof, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IKC123
Record Dates: First submitted 2021-01-13; First posted 2021-01-25 (Actual); Last update posted 2021-01-25 (Actual); Status verified 2021-01

CONDITIONS: Pulmonary Rehabilitation; Lung Cancer
Keywords: pulmonary rehabilitation; lung surgery; lung cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Pulmonary Rehabilitation Group and Control Group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pulmonary Rehabilitation Group (Experimental): An 8-week comprehensive outpatient PR program including respiratory exercises, aerobic and strengthening training
  Interventions: Other: Exercise
- Control Group (Other): Respiratory exercises
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Exercise training

SUMMARY:
Lung cancer is the most common cancer in the world and surgical resection remains the gold standard curative treatment in early stage non-small cell lung cancer. However, surgery itself is the direct cause of pulmonary function impairment, which dramatically reduces patients tolerance to exercise and their quality of life. Pulmonary rehabilitation (PR) complements surgical treatment and improves patients' exercise and functional capacity, decreases dyspnea, improves health status.

Our aim is to examine the effectiveness of PR applied after lung resection in patients with lung cancer, 2- To determine whether the respiratory exercise training given to patients who could not participate in the PR program is effective.

DETAILED DESCRIPTION:
Pulmonary rehabilitation (PR) is an evidence-based, interdisciplinary, comprehensive exercise program that targets patients with symptomatic chronic respiratory disease. PR integrates exercise and training interventions into a personalized treatment program. PR has become an important component of the general treatment strategy in patients with high-risk surgical diseases such as lung resection. It helps patients return to normal not only physically, but also emotionally and mentally. In patients with lung cancer, preoperative PR increases exercise capacity, decreases post-operative morbidity and mortality. Although it is reported that the PR program applied in the post-operative period increases physical performance and improves the quality of life, referral of patients in need of the PR unit is less than 25%. There is a need to increase the awareness of both pulmonologists and thoracic surgeons about the benefits of the PR program, which is a non-pharmacological and effective intervention.

The investigators have had two objectives in this study. 1- To examine the effectiveness of PR applied after lung resection in patients with lung cancer, 2- To determine whether the respiratory exercise training given to patients who could not participate in the PR program is effective.

An 8-week comprehensive outpatient PR program will applied to half of 66 patients with non-small cell lung cancer who underwent lung resection, and the other half received respiratory exercise training. After the intervention, the results of both groups will compare.

ELIGIBILITY:
Inclusion Criteria:

* Patients who had undergone surgery for non-small cell lung cancer in the last two years
* Patients who had no chemotherapy or radiotherapy

Exclusion Criteria:

* Patients who were found unsuitable with the cardiology consultation
* Patients with psychiatric problems
* Patients with severe joint diseases
* Reluctant patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2017-10-01 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Exercise Capacity | up to 8 weeks
  Six minutes walk test

SECONDARY OUTCOMES:
Respiratory Functions | up to 8 weeks
  Pulmonary Function Test Pulmonary function test (PFT) which is noninvasive tests that show how well the lungs are working. The tests will measure FEV1; It is the volume of air (in liters) exhaled in the first second during forced exhalation after maximal inspiration.
  FVC: It s the amount of air that can be forcibly exhaled from your lungs after taking the deepest breath possible, as measured by spirometry FEV1/FVC: It represents the proportion of a person's vital capacity that they are able to expire in the first second of forced expiration (FEV1) to the full, forced vital capacity (FVC).
Dyspnea Sensation | up to 8 weeks
  Modified Medical Research Council (MMRC)" dyspnea scale, which consists of 5 items ranging between 1 and 5, to determine the severity of patients' shortness of breath. Higher scores mean a worse outcome.
Disease Specific Quality of Life | up to 8 weeks
  St. George's Respiratory Questionnaire (SGRQ) to determine disease-specific quality of life. At this scale, high scores define worsened disease and increased symptoms. Higher scores mean a worse outcome.
Anxiety | up to 8 weeks
  Hospital Anxiety and Depression (HAD) Inventory for assessment of anxiety and depression. In this scale; scores of anxiety and depression are calculated separately. The maximum score for both is 21 and high scores correspond to high degree anxiety and depression. Cut-off scores for anxiety and depression were determined as 10/11 and 7/8 respectively.
Depression | up to 8 weeks
  Hospital Anxiety and Depression (HAD) Inventory for assessment of anxiety and depression. In this scale; scores of anxiety and depression are calculated separately. The maximum score for both is 21 and high scores correspond to high degree anxiety and depression. Cut-off scores for anxiety and depression were determined as 10/11 and 7/8 respectively.
Body Mass Index | up to 8 weeks
  Body mass index is calculated by dividing body mass by the square of length in meters

CONTACTS AND LOCATIONS:
Locations (1):
- İlknur Naz Gürşan, Izmir, Turkey (Türkiye)